CLINICAL TRIAL: NCT04901702
Title: A Randomized Phase I/II Study of Talazoparib or Temozolomide in Combination With Onivyde in Children With Recurrent Solid Malignancies and Ewing Sarcoma
Brief Title: Study of Onivyde With Talazoparib or Temozolomide in Children With Recurrent Solid Tumors and Ewing Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Pfizer (Industry); Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONITT; NCI-2021-02843 (Other: NCI)
Record Dates: First submitted 2021-04-30; First posted 2021-05-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Solid Tumor; Recurrent Ewing Sarcoma; Recurrent Hepatoblastoma; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Recurrent Wilms Tumor; Refractory Ewing Sarcoma; Refractory Hepatoblastoma; Refractory Malignant Germ Cell Tumor; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma
Keywords: Pediatric Cancer; Childhood Cancer; Ewing Sarcoma; PARP inhibitor; Solid tumor; Irinotecan; Onivyde; Talazoparib
MeSH Terms: conditions — Sarcoma, Ewing; Hepatoblastoma; Neuroblastoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Wilms Tumor; Neoplasms | interventions — irinotecan sucrosofate; talazoparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (Arm A) ONI plus TAL (Active Comparator): The phase I/II study will evaluate a treatment regimen; nanoliposomal irinotecan (nal-IRN, Onivyde) plus talazoparib (TAL)
  Interventions: Drug: Onivyde; Drug: Talazoparib
- (Arm B) ONI plus TMZ (Active Comparator): The phase I/II study will evaluate a treatment regimen; Onivyde (ONI) plus temozolomide (TMZ)
  Interventions: Drug: Onivyde; Drug: Temozolomide

INTERVENTIONS:
Drug: Onivyde — Given intravenous on Days 1 and 8
  Other Names: Nanoliposomal irinotecan
Drug: Talazoparib — Given orally twice on Day 1 (daily maximum is 1000mcg/day), then daily on Days 2-6
  Other Names: BMN 673; Talzenna
  Arms: (Arm A) ONI plus TAL
Drug: Temozolomide — Given once a day on Days 1-5.
  Other Names: Temodar, Temodal
  Arms: (Arm B) ONI plus TMZ

SUMMARY:
The phase I portion of this study is designed for children or adolescents and young adults (AYA) with a diagnosis of a solid tumor that has recurred (come back after treatment) or is refractory (never completely went away). The trial will test 2 combinations of therapy and participants will be randomly assigned to either Arm A or Arm B. The purpose of the phase I study is to determine the highest tolerable doses of the combinations of treatment given in each Arm.

In Arm A, children and AYAs with recurrent or refractory solid tumors will receive 2 medications called Onivyde and talazoparib. Onivyde works by damaging the DNA of the cancer cell and talazoparib works by blocking the repair of the DNA once the cancer cell is damaged. By damaging the tumor DNA and blocking the repair, the cancer cells may die. In Arm B, children and AYAs with recurrent or refractory solid tumors will receive 2 medications called Onivyde and temozolomide. Both of these medications work by damaging the DNA of the cancer call which may cause the tumor(s) to die.

Once the highest doses are reached in Arm A and Arm B, then "expansion Arms" will open. An expansion arm treats more children and AYAs with recurrent or refractory solid tumors at the highest doses achieved in the phase I study. The goal of the expansion arms is to see if the tumors go away in children and AYAs with recurrent or refractory solid tumors. There will be 3 "expansion Arms". In Arm A1, children and AYAs with recurrent or refractory solid tumors (excluding Ewing sarcoma) will receive Onivyde and talazoparib. In Arm A2, children and AYAs with recurrent or refractory solid tumors, whose tumors have a problem with repairing DNA (identified by their doctor), will receive Onivyde and talazoparib. In Arm B1, children and AYAs with recurrent or refractory solid tumors (excluding Ewing sarcoma) will receive Onivyde and temozolomide.

Once the highest doses of medications used in Arm A and Arm B are determined, then a phase II study will open for children or young adults with Ewing sarcoma that has recurred or is refractory following treatment received after the initial diagnosis. The trial will test the same 2 combinations of therapy in Arm A and Arm B. In the phase II, a participant with Ewing sarcoma will be randomly assigned to receive the treatment given on either Arm A or Arm B.

DETAILED DESCRIPTION:
ONITT (ONIvyde, Talazoparib, Temozolomide) is a phase I/II study which will evaluate two treatment regimens; nanoliposomal irinotecan (nal-IRN, Onivyde) plus talazoparib (TAL) and Onivyde (ONI) plus temozolomide (TMZ) for the treatment of recurrent or refractory (RR) Ewing sarcoma. A dose finding phase I study will be open to patients with recurrent or refractory solid tumors. Patients will be assigned to receive either ONI plus TAL (Arm A) or ONI plus TMZ (Arm B). Once the recommended phase II doses (RP2D) of Arm A and Arm B are determined, expansion cohorts (A1, B1) will open at the RP2Ds for enrollment of non-Ewing sarcoma solid tumor patients. There will be an additional Arm A expansion cohort (A2) for patients with homologous recombination repair defects. Concurrently, the phase II study will open to patients with RR Ewing sarcoma. In the phase II study, patients with RR Ewing sarcoma will be randomized to receive either ONI plus TAL or ONI plus TMZ. The primary endpoint will be progression-free survival (PFS). PFS of both treatment arms in the phase II study will be compared to one another by using a two-arm non-inferiority design when superiority is expected.

Phase I Primary Objective To determine the recommended phase 2 doses (RP2Ds) of Onivyde combined with talazoparib (Arm A) and Onivyde combined with temozolomide (Arm B) administered to children, adolescents and young adults with refractory or recurrent solid malignancies.

Phase I Secondary Objectives

* To characterize the safety profile of the drug regimens, Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B).
* To characterize the plasma pharmacokinetics (PK) of Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent solid malignancies.
* To estimate the antitumor activity of Onivyde plus talazoparib and Onivyde plus temozolomide.

Phase I Exploratory Objectives

* To describe the relationship between UGT1A1 genotype status with toxicity and response.
* To describe the molecular germline and somatic profiles, including evaluation of mutations in homologous recombination genes and their possible association to therapy response in participants with recurrent or refractory solid tumors.
* To measure ctDNA at different time points and evaluate its relationship with response to therapy.
* To describe the safety of onivyde plus talazoparib vs onivyde plus temozolomide at the determined RP2D in children, adolescents and young adults treated in the expansion cohorts.
* To describe the palatability and ease of administration of talazoparib liquid suspension in children who are unable to swallow the capsules.

Phase II Primary Objectives

• To compare the progression-free survival (PFS) of Onivyde plus talazoparib and Onivyde plus temozolomide in participants with refractory or recurrent Ewing sarcoma.

Phase II Secondary Objectives

* To describe the toxicity of the treatment regimens.
* To describe the objective response rate (ORR), disease control rate (DCR) after cycle 4, duration of response (DoR), event free survival (EFS) and overall survival (OS) for participants receiving Onivyde plus talazoparib and Onivyde plus temozolomide.
* To characterize the plasma pharmacokinetics of Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma.

Phase II Exploratory Objectives

* To describe the relationship between UGT1A1 genotype status with toxicity and response.
* To describe the molecular germline and somatic profiles, including evaluation of mutations in homologous recombination genes and their possible association to chemotherapy response in participants with recurrent or refractory Ewing sarcoma.
* To describe ctDNA at different time points and the relationship with response to therapy.
* To describe the palatability and ease of administration of talazoparib liquid suspension in children who are unable to swallow the capsules.

Phase I The phase I portion of the study will include 2 separate treatment arms, Arms A and B. Arm A will evaluate Onivyde plus talazoparib (ONI + TAL). Arm B will evaluate Onivyde plus temozolomide (ONI + TMZ). Both phase I studies will be open to patients with recurrent or refractory solid tumors who meet eligibility criteria. In Arm A, patients will receive intravenous Onivyde on Days 1 and 8. They will receive oral talazoparib twice on Day 1 and then daily on Days 2-6. In Arm B, participants will receive intravenous Onivyde on Days 1 and 8. They will receive oral temozolomide daily on Days 1-5. Pharmacokinetic testing will take place during Cycle 1. Therapy may continue for up to 24 months. Tumor assessments will be performed at baseline and repeated after cycles 2, 4, 6 and then every 4 cycles thereafter to assess disease status. If at any designated disease evaluation time point a patient develops a response that is better than the prior response (i.e. SD at Cycle 2 evaluation, then PR at Cycle 4 evaluation), an interim disease evaluation is recommended after 28 days to confirm response. Therapy will be discontinued if there is evidence of disease progression or drug-related dose limiting toxicities requiring removal from treatment. Safety and tolerability will be monitored continuously throughout study participation.

Phase II Following the completion of the phase I dose finding studies, patients with recurrent or refractory Ewing sarcoma that meet eligibility criteria will be eligible for randomization into the phase II study. Arm A will evaluate Onivyde plus talazoparib (ONI + TAL). Arm B will evaluate Onivyde plus temozolomide (ONI + TMZ). In Arm A, patients will receive intravenous Onivyde on Days 1 and 8. They will receive oral talazoparib twice on Day 1 and then daily on Days 2-6. In Arm B, patients will receive intravenous Onivyde on Days 1 and 8. They will receive oral temozolomide daily on Days 1-5. Pharmacokinetic testing will take place during Cycle 1. Therapy may continue for up to 24 months. Tumor assessments will be performed at baseline and repeated after Cycles 2, 4, 6 and then every 4 cycles thereafter to assess disease status. If at any designated disease evaluation time point a patient develops a response that is better than the prior response (i.e. SD at Cycle 2 evaluation, then PR at Cycle 4 evaluation), an interim disease evaluation is recommended after 28 days to confirm response. Therapy will be discontinued if there is evidence of disease progression and/or any other condition(s) occur that do not allow treatment continuation or similar toxicities requiring removal from the trial. Safety and tolerability will be monitored continuously throughout study participation.

Sample size: In the dose escalation phase I study, approximately 18 patients per arm will be enrolled for a total of 36 patients. The dose expansion phase I study will include 3 treatment cohorts. Arm A will have 2 dose expansion cohorts including 1) a non-ES solid tumor cohort (A1) and 2) a DNA repair defects/mutations cohort (A2). Arm B will have 1 dose expansion cohort including non-ES solid tumors (B1). Approximately 12 patients will enroll per expansion treatment cohort for a total of 36 patients. In the phase II study, 44 patients will be enrolled on each arm for a total of 88 patients.

ELIGIBILITY:
Inclusion Criteria

Patients must be > 12 months and < 30 years at the time of enrollment on study.

Phase I

* Patients with refractory or recurrent non-central nervous system (CNS) solid tumors not amenable to curative treatment are eligible. Patients must have had histologic verification of malignancy at original diagnosis or at the time of relapse. Patients eligible for the expansion cohort, A2, will include non-ES patients with refractory or recurrent non-CNS solid tumors with a deleterious alteration in germline or somatic genes involved in HR repair and DSBs signaling, germline or somatic assessed by prior comprehensive sequencing performed in a CLIA-approved (or equivalent) facility.

Phase II

* Patients with refractory or recurrent Ewing sarcoma (during or after completion of first-line therapy). Refractory disease is defined as progression during first line treatment or within 12 weeks of completion of first line treatment. Recurrent disease includes patients who received first line treatment and experienced disease progression at any time point >12 weeks from the completion of first line therapy.
* Patients must have a histologic diagnosis of Ewing sarcoma with EWSR1- FLI1 translocation or other EWS rearrangement at the time of initial diagnosis. Repeat biopsy at the time of disease recurrence is strongly encouraged but it is not required/mandated for enrollment.

Disease status

* Patients must have either measurable or evaluable disease (see Section 7.0 for definitions). Measurable disease includes soft tissue disease evaluable by cross-sectional imaging (RECIST). Patients with bone disease without a measurable soft tissue component or bone marrow disease only are eligible for the phase 1 and phase 2 study but will not be included in the OR endpoint.
* Performance level: Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients < 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior therapy

Phase I Patients who have received prior therapy with an irinotecan-based or temozolomide-based regimen are eligible. Patients who have received prior therapy with a PARP inhibitor other than talazoparib are eligible.

Phase II

* Patients should have received first line therapy and developed either refractory or recurrent disease (first relapse).
* Organ function: Must have adequate organ and bone marrow function as defined by the following parameters:
* Patients with solid tumors not metastatic to bone marrow:
* Peripheral absolute neutrophil count (ANC) >1,000/mm3 (1x109/L)
* Platelet count > 75,000/mm3 (75x109/L) (no transfusion within 7 days of enrollment)
* Hemoglobin > 9 g/dL (with or without support)

In the phase I study, patients with solid tumors metastatic to bone marrow or with bone marrow hypocellularity defined as <30% cellularity in at least one bone marrow site will be eligible for study, but they will not be evaluable for hematologic toxicity. These patients must not be refractory to red cell or platelet transfusions. At least 2 of every cohort of 3 patients (in the phase I study) must be evaluable for hematologic toxicity. If dose limiting hematologic toxicity is observed at any dose level, all subsequent patients enrolled at that dose level must be evaluable for hematologic toxicity.

* Adequate renal function defined as: Creatinine clearance or radioisotope GFR > 60ml/min/1.73m2 or a serum creatinine maximum based on age/sex: age 6months to <1 year, creatinine 0.4; 1 to < 2 years, creatinine 0.6; 2 < 6 years, creatinine 0.8; 6 < 10 years, creatinine 1; 10 to <13 years, creatinine 1.2; 13 to < 16 years creatinine 1.5 (males) or 1.4 (females); > 16 years, creatinine 1.7 (males) 1.4 (females)
* Adequate liver function defined as: normal liver function as defined by SGPT (ALT) concentration <5x the institutional ULN, a total bilirubin concentration <2x the institutional ULN for age, and serum albumin > 2g/dL.
* Adequate pulmonary function defined as no evidence of dyspnea at rest and a pulse oximetry > 94% if there is a clinical indication for determination. Pulmonary function tests are not required.
* Patients must have fully recovered from the acute toxic effects of chemotherapy, immunotherapy, surgery, or radiotherapy prior to entering this study:
* Myelosuppressive chemotherapy: Patient has not received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (8 weeks if received prior myeloablative therapy).
* Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim.
* Biologic (anti-neoplastic agent): At least 7 days must have elapsed since completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur.
* Monoclonal antibodies: At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody or 28 days have elapsed since last dose of the monoclonal antibody with complete resolution of symptoms related to treatment.
* Radiotherapy: At least 2 weeks must have elapsed since any irradiation; at least 6 weeks must have elapsed since craniospinal RT, 131I-mIBG therapy or substantial bone marrow irradiation (e.g., >50% pelvis irradiation).
* Female participant who is post-menarchal must have a negative urine or serum pregnancy test and must be willing to have additional serum and urine pregnancy tests during the study.
* Female or male participant of reproductive potential must agree to use effective contraceptive methods at screening and throughout duration of study treatment.

Exclusion Criteria

Pregnant or breastfeeding

* Pregnant or breast-feeding women will not be entered on this study. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two methods of birth control: a medically accepted barrier of contraceptive method (e.g., male or female condom) and a second method of birth control during protocol therapy. Two highly effective methods of contraception are required for female patients during treatment and for at least 7 months after completing therapy. Male patients with female partners of reproductive potential and/or pregnant partners are advised to use two highly effective methods of contraception during treatment and for at least 4 months after the final dose.
* Male and female participants must agree not to donate sperm or eggs, respectively, after the first dose of study drug through 105 days and 45 days after the last dose of study drug. Females considered not of childbearing potential include those who are surgically sterile (bilateral salpingectomy, bilateral oophorectomy, or hysterectomy).

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I:To determine the recommended phase 2 doses (RP2Ds) of Onivyde combined with talazoparib (Arm A) and Onivyde combined with temozolomide (Arm B) administered to children, adolescents and young adults with refractory or recurrent solid malignancies. | approximately 21 days
  First cycle dose limiting toxicity (DLTs) will be used to determine the RP2Ds of the two treatment arms. The DLT is defined as any of the following events that are possibly, probably or definitely attributable to protocol therapy.
Phase II:To estimate the progression-free survival (PFS) of Onivyde plus talazoparib and Onivyde plus temozolomide in patients with refractory or recurrent Ewing sarcoma. | for five years following the date the last patient was randomized
  The study is designed to compare the progression-free survival (PFS) of Onivyde plus talazoparib and Onivyde plus temozolomide in patients with refractory or recurrent Ewing sarcoma. PFS is defined as the time from randomization to disease progression or death, whichever is earlier.

SECONDARY OUTCOMES:
Phase I:To characterize the safety profile of the treatment regimens, Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment (up to 24 months after enrollment of last participant)]
  Safety and tolerability will consist of monitoring and recording all AEs and SAEs as characterized by type, frequency, severity, timing, seriousness and the relationship to the study therapy. These will be reported out qualitatively.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: maximum plasma concentration (Cmax) on Day 1 and Day 6; for Onivyde: maximum plasma concentration (Cmax) on Day 1 .
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: Tmax on Day 1 and Day 6; for Onivyde: Tmax on Day 1 .
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For both talazoparib and Onivyde: clearance (CL) in Cycle 1.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: area under the plasma concentration time curve (AUCtau (AUC24)) in Cycle 1.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: Ctrough (predose) in Cycle 1.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For Onivyde: area under the plasma concentration time curve (AUCinf) in Cycle 1.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For Onivyde: half-life (t½) on Day 1.
To characterize the plasma pharmacokinetics of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided For Onivyde: Vd on Day 1.
To estimate the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At time of randomization until evaluation of respective endpoints, up to 4 months after enrollment of last participant
  Descriptive statistics of objective response rate (ORR) at cycle 4 will be provided.
To estimate the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At time of randomization until evaluation of respective endpoints, up to 4 months after enrollment of last participant
  Descriptive statistics of disease control rate (DCR) at cycle 4 will be provided.
To estimate the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At time of randomization until evaluation of respective endpoints up to 4 months after enrollment of last participant
  Descriptive statistics of duration of response (DoR) will be provided.
To estimate the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At time of randomization until evaluation of respective endpoints, up to 2 years after enrollment of last participant
  Descriptive statistics event-free survival (EFS) will be provided.
To estimate the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At time of randomization until evaluation of respective endpoints, up to 2 years after enrollment of last participant
  Descriptive statistics of overall survival (OS) will be provided.
Phase II: To describe the toxicity of the treatment regimens. | At the end of treatment (up to 24 months after enrollment of last participant)
  Safety and tolerability will consist of monitoring and recording all AEs and SAEs as characterized by type, frequency, severity, timing, seriousness and the relationship to the study therapy. These will be reported out qualitatively.
To describe the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment, up to 24 months after enrollment of last participant
  Descriptive statistics of objective response rate (ORR) at cycle 4 will be provided.
To describe the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment, up to 24 months after enrollment of last participant
  Descriptive statistics of disease control rate (DCR) at cycle 4 will be provided.
To describe the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment, up to 24 months after enrollment of last participant
  Descriptive statistics of duration of response (DoR) will be provided.
To describe the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment, up to 5 years after randomization of last participant
  Descriptive statistics of event-free survival (EFS) will be provided.
To describe the antitumor activity of Onivyde plus talazoparib (Arm A) and Onivyde plus temozolomide (Arm B) | At the end of treatment, up to 5 years after randomization of last participant
  Descriptive statistics of overall survival (OS) will be provided.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: maximum plasma concentration (Cmax) on Day 1 and Day 6; for Onivyde: maximum plasma concentration (Cmax) on Day 1 .
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: Tmax on Day 1 and Day 6; for Onivyde: Tmax on Day 1 .
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of cycle 1 (approximately 21 days after last participant enrollment
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For both talazoparib and Onivyde: clearance (CL) in Cycle 1.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: area under the plasma concentration time curve (AUCtau (AUC24)) in Cycle 1.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For talazoparib: Ctrough (predose) in Cycle 1.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma | At the end of cycle 1 (approximately 21 days after last participant enrollment)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For Onivyde: area under the plasma concentration time curve (AUCinf) in Cycle 1.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided. For Onivyde: half-life (t½) on Day 1.
To characterize the plasma pharmacokinetics Onivyde and talazoparib in children, adolescents and young adults with refractory or recurrent Ewing sarcoma. | At the end of Cycle 1 (each cycle is 21 days)
  Descriptive statistics of plasma drug concentrations and pharmacokinetic parameters will be provided For Onivyde: Vd on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (10):
- United States (7):
  - Lucille Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta/Emory University School of Medicine, Atlanta, Georgia
  - Children's Hospital and Clinics of Minn, Minneapolis, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital/ Baylor College of Medicine, Houston, Texas
- Canada (3):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal
  - BC Children's Hospital Research Institute, Vancouver

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols